CLINICAL TRIAL: NCT04229602
Title: Bioequivalence Study of Venlafaxine Hydrochloride Sustained-Release Capsules and EFEXOR® XR Under Fed Conditions in Chinese Healthy Volunteers
Brief Title: Bioequivalence Study of Venlafaxine Hydrochloride Sustained-Release Capsules in Chinese Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FY-CP-06-201909-01
Record Dates: First submitted 2019-12-31; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Bioequivalence Study
MeSH Terms: interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venlafaxine Hydrochloride Sustained-Release Capsules (Experimental): During the study session, healthy subjects will be administered a single dose of Hydrochloride Sustained-Release Capsules 75 mg under Fed conditions.
  Interventions: Drug: Venlafaxine Hydrochloride Sustained-Release Capsules 75 mg
- Active Comparator: EFEXOR® XR (Active Comparator): During the study session, healthy subjects will be administered a single dose of EFEXOR® XR 75mg under Fed conditions.
  Interventions: Drug: EFEXOR® XR

INTERVENTIONS:
Drug: Venlafaxine Hydrochloride Sustained-Release Capsules 75 mg — A generic product manufactured by Beijing Winsunny Pharmaceutical Co., Ltd.
  Arms: Venlafaxine Hydrochloride Sustained-Release Capsules
Drug: EFEXOR® XR — EFEXOR® XR (75mg) produced by Pfizer Ireland Pharmaceuticals(held by Pfizer Healthcare Ireland, distributed by Wyeth pharmaceutical co. LTD)
  Arms: Active Comparator: EFEXOR® XR

SUMMARY:
The objective of this study is to evaluate the human bioequivalence of two Venlafaxine Hydrochloride Sustained-Release Capsules (75 mg) .

DETAILED DESCRIPTION:
The objective of this study is to evaluate the human bioequivalence of Venlafaxine Hydrochloride Sustained-Release Capsules (75 mg) produced by Beijing Winsunny Pharmaceutical Co., Ltd and EFEXOR® XR (75mg) produced by Pfizer Ireland Pharmaceuticals(held by Pfizer Healthcare Ireland, distributed by Wyeth pharmaceutical co. LTD), as well as the safety of the tested preparation, and to provide basis for the evaluation of the quality and efficacy consistency of the tested preparation and the reference preparation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are fully informed and voluntarily consent to participate in this study;
2. Healthy adult volunteers of ≥18 years old and ≤ 65 years old, male or female;
3. Body weight ≥ 50.0 kg for male and 45.0 kg for female;
4. Subjects are able to communicate well with the investigator and to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Subjects enroll in other clinical trials and take corresponding experimental drugs within 90 days before the trial, or participate in other clinical trials;
2. The results of physical examination, vital signs examination, clinical laboratory examination (blood routine, urine routine, blood biochemistry, coagulation function, immunity 8 items, blood pregnancy (female only)), 12-lead electrocardiogram (ECG) are clinical significant;
3. Any previous history and present medical history that may affect the safety of the trial or the in-vivo process of the drug, especially a history of liver, kidney, endocrine, cardiovascular, nervous, gastrointestinal, lung, tumor, immune, skin, blood or metabolic disorders that the investigator considers clinically significant;
4. Any history of surgery or trauma that may affect the safety of the test or the in-vivo process of the drug;;
5. Subjects have depression, mania and other mental disorders, or have suicidal tendencies;
6. Subjects have the history of angle-closure glaucoma;
7. Heavy smokers (average daily smoking of more than 5 cigarettes in the 90 days before the trial), heavy drinkers (average weekly drinking of more than 14 units of alcohol in the 90 days before the trial, 1 unit =360 mL beer or 45 mL 40% spirits or 150 mL wine), and subjects who could not promise to quit smoking and drinking during the experiment;
8. Subjects had taken any alcoholic product within 24 hours before the test, or had tested positive for alcohol breath test;
9. Allergic to any component of venlafaxine hydrochloride sustained-release capsules, or with a history of specific allergies (asthma, urticaria, eczema, etc.), or allergic constitution (such as allergic to two or more drugs or food);
10. Lactose intolerance (a history of diarrhea from drinking milk);
11. Previous history of drug use, drug abuse, or positive urine drug screening;
12. Subjects who have donated blood or lost blood equal to or more than 200 mL within 90 days before the test, received blood transfusion or used blood products, or intend to donate blood or blood components during or within 3 months after the test;
13. Nursing woman;
14. Subjects planned parenthood, unwillingness or inability to use effective contraception, within 30 days before the trial (for women), and within six months after the end of the trial;
15. Subjects who have taken any medicine (including Chinese herbal medicine) and health care products within 14 days before the test;
16. Subjects who have taken any medicine that interacts with the drug or alters liver enzyme activity within 30 days prior to the trial, such as cimetidine, haloperidol, ketoconazole, clot-disrupting drugs (such as non-steroidal anti-inflammatory drugs, aspirin and warfarin), Monoamine oxidase inhibitors (such as phenyledrine, phenylamine, isazolid, isazolid, moclobemide, bromofaramine, nyalamide, tloxadone, defloxadone, slegiline, linezolid, or methylene blue for intravenous use), similar to other serotonin drugs (including triptans, selective serotonin reuptake inhibitors (SSRIs), other serotonin and norepinephrine reuptake inhibitors (SNRIs), lithium, sibutramine, tramadol or st John's wort, and tryptophan supplements) etc ;
17. Subjects who have eaten special diet (including grapefruit and/or food or drink rich in xanthine derivatives or alcohol, such as tea and coffee, etc.) or have other factors affecting drug absorption, distribution, metabolism and excretion within 14 days before the test;
18. Subjects who have special requirements on diet and cannot accept unified diet;
19. Subjects who have the difficulty in venous blood, or can not tolerate venipuncture, or have a history of dizziness;
20. Subjects who need to drive and operate machines or engage in other potentially dangerous activities during the test;
21. Other situations that the researchers considered unsuitable to enroll the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-04-02 (Estimated); Study Completion 2020-07-02 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax | Blood samples collected over 72 hour period
  Cmax - Maximum Observed Concentration (of Venlafaxine in Plasma)
Bioequivalence based on AUC0-t | Blood samples collected over 72 hour period
  AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Bioequivalence based on AUC0-∞ | Blood samples collected over 72 hour period
  AUC0-∞- Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zhao, Dr, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Institution of Drug Clinical Trials, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No